CLINICAL TRIAL: NCT06595043
Title: Effects of Different Occlusion Angles of Disposable Tracheal Blocker on Right One-lung Ventilation: a Multi-center, Prospective, Randomized Controlled Trial
Brief Title: Effects of Different Occlusion Angles of Disposable Tracheal Blocker on Right One-lung Ventilation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University, China (Other)
Responsible Party: Principal Investigator, Wenfei Tan, Professor,Chairman, China Medical University, China
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20240910
Record Dates: First submitted 2024-09-09; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: The Direction of Blocker Placement

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the tip opening angle to the left (Experimental): After fixing the position of the tracheal catheter, the opening of the tip of the blocker will be adjusted to left under the guidance of the fiber bronchoscope.
  Interventions: Device: the tip opening angle to the left
- the tip opening angle to the right (Placebo Comparator): After fixing the position of the tracheal catheter, the opening of the tip of the blocker will be adjusted to right under the guidance of the fiber bronchoscope.
  Interventions: Device: the tip opening angle to the right

INTERVENTIONS:
Device: the tip opening angle to the left — After fixing the position of the tracheal catheter, the opening of the tip of the blocker will be adjusted to left under the guidance of the fiber bronchoscope.
  Arms: the tip opening angle to the left
Device: the tip opening angle to the right — After fixing the position of the tracheal catheter, the opening of the tip of the blocker will be adjusted to right under the guidance of the fiber bronchoscope.
  Arms: the tip opening angle to the right

SUMMARY:
This trial is a practical, multicenter, prospective, parallel grouping, randomized controlled,two-arm study. This study will be conducted in three centers including the First Hospital of China Medical University, Seoul National University Hospital and the University Clinical Center of Serbia. The investigators aim to investigate the effect of different occlusion angles of disposable tracheal blocker on right one-lung ventilation

DETAILED DESCRIPTION:
This trial is a practical, multi-center, prospective, parallel grouping, randomized controlled,two-arm clinical study comparing the different occlusion angles of disposable tracheal blocker on right one-lung ventilation. It is planned to enroll 96 subjects requiring right-sided One-Lung ventilation, aged 18-65 years, at three centers. Patients will be randomly assigned to the tip opening angle to the right (Group R), or he tip opening angle to the left (Group L). The primary outcome is the satisfaction with intraoperative collapse of the right lung. The secondary outcome is the one-time success rate of occuder implantation

ELIGIBILITY:
Inclusion Criteria:

* Age ranged from 18 to 65 years old;
* American Society of Anesthesiologists (ASA) grade I-III;
* No history of drug allergy or abnormal anesthesia;
* Patients undergoing right thoracoscopic surgery;
* The preoperative oxygen saturation was not less than 94%.

Exclusion Criteria:

* Patients with a history of acute lung injury or ARDS within 3 months;
* Cardiac function class IV (New York Heart Association classification);
* Chronic renal failure (renal cell filtration rate <30ml min-11.73m-2), severe liver disease;
* Patients with blurred consciousness and cognitive dysfunction;
* Patients with severe coagulation dysfunction;
* Without preoperative oxygen inhalation, blood oxygen <94%, severe pulmonary dysfunction;
* Patients with endotracheal tube admitted to ICU after operation;
* Body mass index (BMI) >30;
* Patients who had had lung surgery；
* Inability to complete the study;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2024-10-09 (Estimated); Primary Completion 2025-10-09 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Satisfaction with the collapse of the right lung | On the 3 minutes after one lung ventilation
  The pirimary outcome is the comparison the effects of different occluder opening directions on lung collapse by one surgeon using lung collapse score (1-4, 4 means the best)

SECONDARY OUTCOMES:
The first time success rate of blocker implantation | On the time of blocker implantation 30 seconds
  The first time success rate of blocker implantation

CONTACTS AND LOCATIONS:
Locations (3):
- Wenfei Tan, Shenyang, China
- the University Clinical Center of Serbia, Belgrade, Serbia
- Konkuk University School of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR
Time Frame: On the time of paper published